CLINICAL TRIAL: NCT02090543
Title: Rivaroxaban Versus Vitamin K-Antagonist (VKA) in Thromboprophylaxis of Patients With Atrial Fibrillation: Patient Preference Study
Brief Title: BAY 59-7939 (Xarelto, SPAF), Non Interventional Studies
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 17019; OR-ITW-01-13 (Other: Company internal)
Record Dates: First submitted 2014-02-12; First posted 2014-03-18 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Phenprocoumon; Rivaroxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: 300 AF patients, with at least 3 month of anticoagulation therapy with VKAs (VKA-experienced patients)
  Interventions: Drug: Phenprocoumon (Marcumar)
- Group 2: 300 AF patients, with at least 3 month of rivaroxaban therapy (rivaroxaban-experienced patients)
  Interventions: Drug: Rivaroxaban (Xarelto, BAY-59 7939)

INTERVENTIONS:
Drug: Phenprocoumon (Marcumar) — common use, no requirements (real life situation)
  Groups: Group 1
Drug: Rivaroxaban (Xarelto, BAY-59 7939) — common use, no requirements (real life situation)
  Groups: Group 2

SUMMARY:
According to recent guidelines, long-term anticoagulation is recommended for patients with atrial fibrillation (AF) and a risk profile with CHA2DS2-VASc score of 1 or more. Vitamin K antagonists(VAK) and novel oral anticoagulants such as rivaroxaban are current treatment options for AF patients with additional risk factors for stroke. Currently there are only limited information to what extend AF patients prefer one or the other treatment option based on patient relevant characteristics of novel oral anticoagulants vs. VKAs. It is also unknown which of the characteristics influences patient preference most and how this relates to a neutral comparator. Furthermore, an additional unknown factor is also how patient evaluate their current treatment and if this leads to differences among treatment with VKAs and rivaroxaban.

ELIGIBILITY:
Inclusion Criteria:

A.General Criteria (Group 1and Group2):

* diagnosed non-valvular AF
* older than 18 years
* general capability and willingness to perform a structured patient interview in German
* no participation in any other clinical or observational study over the last 3 month

Additional criteria for Group1 (VKA-experienced):

* active VKA-therapy for at least 3 month without significant interruptions
* in case of perioperative interruption VKA treatment should not have been hold for more than two weeks.

Additional criteria for Group2 (rivaroxaban-experienced patients):

* active rivaroxaban-therapy for at least 3 month without significant interruptions
* in case of perioperative interruption VKA treatment should not have been hold for more than two weeks.

Exclusion Criteria:

* participation in any other clinical or observational study over the last 3 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult AF-patients, within 3 month of anticoagulation (VKA or rivaroxaban) therapy, recruited by GPs
Sampling Method: Non-Probability Sample
Enrollment: 647 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
A prescription of patient preferences pattern including 5 attributes for Discrete-Choice-Experiment(DCE)-design in patients with atrial fibrillation | Within 1-4 weeks after patient enrollement
  Attributes and values in relation to the DCE-Choice-Set. The patient will receive a "test card" with the following attributes: bridging of anticoagulation, regular anticoagulation control, limitations to eating behaviour and alcohol consumption, once vs. twice daily intake of medication, neutral comparator for quantification display of preference: distance to therapy practice
Patient relevant burden/benefit due to anticoagulation using the ACTS-questionnaire | At study entry

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Germany